CLINICAL TRIAL: NCT06155097
Title: Role of Transversus Thoracis Plane Block Versus Parasternal Intercostal Nerve Plane Block in Enhanced Recovery Program After Cardiac Surgery: A Randomized Controlled Study
Brief Title: Transversus Thoracis Plane Block Versus Parasternal Intercostal Nerve Plane Block for Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rehab Abd-Allah Wahdan, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-11-2023
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Surgery
Keywords: postcardiac surgery; transversus thoracis muscle plane block; parasternal intercostal nerve block; Enhanced recovery after surgery

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 3 groups by a computer-generated randomization table
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded (patient and outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Patients will not receive any regional injections
- The transversus thoracis muscle plane block (TTP) group (Active Comparator): Patients will receive the TTP block with administration of 20 ml volume of local anesthetics (Lidocaine 2% + Bupivicaine 0.5% 1:1 mixture + 8mg dexamethasone) bilaterally
  Interventions: Drug: transversus thoracis muscle plane block (TTP)
- The parasternal intercostal nerve block (PSI block) group (Active Comparator): Patients will receive the PSI block with administration of 20 ml volume of local anesthetics (Lidocaine 2% + Bupivicaine 0.5% 1:1 mixture + 8mg dexamethasone) bilaterally
  Interventions: Drug: parasternal intercostal nerve block (PSI block)

INTERVENTIONS:
Drug: transversus thoracis muscle plane block (TTP) — patient in supine position with chest exposed and monitored by beat-to-beat arterial tracing and standard monitors. After determining the anterior T4-T5 interspace using US, the US probe places in the longitudinal plane 1 cm lateral to the sternal border. A parasternal sagittal view of the internal intercostal muscle and the transversus thoracis muscle between the fourth and fifth rib will be visualized above the pleura. A 22-gage needle will be inserted in plane to the transducer with the tip of the needle located in the TTP between the internal intercostal and transversus thoracis muscles. After excluding intravascular and intrapleural placement, LA will administer with intermittent aspiration (administration of 20 ml volume of local anesthetics (Lidocaine 2% +Bupivicaine 0.5% 1:1 mixture + 8mg dexamethasone) on each side. After block administration, the patients will be monitored for LA toxicity, hemodynamic instability, and allergic or unexpected adverse reactions for 20 minutes.
  Arms: The transversus thoracis muscle plane block (TTP) group
Drug: parasternal intercostal nerve block (PSI block) — patient in supine position with chest exposed and monitored by beat-to-beat arterial tracing and standard. Ultrasound scan will be performed from lateral to medial in the intercostal space. The intercostal muscles and pleura will be identified along the lower border of the rib. At the lateral border of the sternum, internal thoracic vessels lying anterior to transverse thoracic muscle are identified. The needle will be inserted in-plane to follow its tip using 4-mL injections per intercostal space across levels two through six bilaterally, for a total of 40 mL (Lidocaine 2% +Bupivicaine 0.5% 1:1 mixture + 8mg dexamethasone)
  Arms: The parasternal intercostal nerve block (PSI block) group

SUMMARY:
Traditionally postoperative pain management after cardiac surgery has been based on opiate analgesics. However, opiates have some undesirable dose-related side-effects such as nausea, constipation, vomiting, dizziness, mental confusion and respiratory depression, which substantially influence patient recovery and may delay discharge after surgery.

The American Society of Anesthesiologists has endorsed multi- modal analgesia, involving multiple analgesics with differing modes of action, to reduce the overreliance on opioid-based postsurgical analgesic regimens and the associated adverse effects.

The safety of using the transversus thoracis muscle plane block (TTP) or the parasternal intercostal nerve block (PSI block) for cardiac surgeries allow to make the option of using opioids alone and the possibility of its complications not the rule in post-operative pain relief in cardiac surgeries.

In the current study, improving the quality of the transversus thoracis muscle plane block (TTP) or the parasternal intercostal nerve block (PSI block) for cardiothoracic surgeries by enhancing post-operative pain relief becomes more and more required to cope up with the new surgical modalities.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) is an international effort to develop perioperative programs aimed at optimizing patient outcomes and healthcare delivery efficiency. These programs are composed of intervention bundles based on the principles of best practice, standardized and consistent healthcare delivery, regular audit, and team feedback, all with a patient-centered focus. Implementation of such programs has resulted in patient and healthcare benefits, including promising early results within the cardiac surgical community.

A perioperative, multimodal, opioid-sparing, pain management plan is classified as B-NR (B-level evidence, nonrandomized studies) in the classification of recommendation and level of evidence. The ERAS Cardiac Society's grading of this recommendation is appropriate because it is a laudable goal that requires additional research. Areas of investigation to refine postoperative pain management include the following: managing patient and provider expectations, individualizing the dose and types of analgesics, consideration of the potential cardioprotective effects of opioids, and incorporating nonpharmacologic approaches to pain management such as regional anesthesia.

Pain after cardiac surgery is caused by several factors; sternotomy, sternal/rib retraction, pericardiotomy, internal mammarian artery harvesting, saphenous vein harvesting, surgical manipulation of the parietal pleura, chest tube insertion and other musculoskeletal trauma during surgery.

Postoperative pain management remains an important clinical challenge in cardiothoracic surgery. Inadequate postoperative pain control may have adverse pathophysiologic sequelae, including increased myocardial oxygen demand, hypoventilation, suboptimal clearance of pulmonary secretions, acute respiratory failure, and decreased mobility, with associated increased risks for thromboembolic events. These adverse events may result in greater perioperative morbidity and mortality.

Despite several multimodal approaches to postoperative pain control, optimal pain management after cardiothoracic procedures remains elusive.

Regional anesthesia (RA) is often included in enhanced recovery protocols (ERPs) as an important component of a bundle of interventions to improve outcomes after surgery. Regional anesthesia techniques, including neuraxial and peripheral nerve block, can provide many benefits for patients in the perioperative period. These benefits include a decrease in postoperative pain (subsequently reducing opioid consumption and associated adverse effects), decrease in nausea and vomiting, improvement in mobilization and recovery of gastrointestinal function, decrease in length of stay (LOS), reduction in surgical stress response, and potentially, reduction in morbidity and mortality. They are therefore commonly used to improve quality of patient care and have also been used as a key component of many enhanced recovery protocols (ERPs).

The transversus thoracis muscle plane block (TTP) is a newly developed regional anesthesia technique which provides analgesia to the anterior chest wall. First described by Ueshima and Kitamura in 2015, the TTP block is a single-shot nerve block that deposits local anesthetic in the transversus thoracis muscle plane between the internal intercostal and transversus thoracis muscles. In the original ultrasound- guided cadaveric study, the TTP block was found to cover the T2-T6 intercostal nerves.

The anterior branches of these intercostal nerves dominate the sensory innervation of the internal mammary region, suggesting this new technique had potential to provide analgesia for surgery of the anterior chest wall.

Another technique for blocking multiple anterior branches of intercostal nerves, named the parasternal intercostal nerve block (PSI block). To perform a PSI block, we inject a local anesthetic between the pectoral major muscle and the external intercostal muscle. Because anterior branches of the intercostal nerve penetrate through these two muscles to innervate the internal mammary area, injection of a local anesthetic to this plane could block anterior branches of intercostal nerves.

Parasternal intercostal nerve blocks using local anesthetic agents have been shown to provide improved postoperative pain control and decreased opioid requirements with fewer potential complications.

This study can reduce economic cost by ENHANCED RECOVERY After Surgery (ERAS) (early extubation, reduce ICU and hospital stay) and improving postoperative analgesia. Implementation of such programs has resulted in patient and healthcare benefits, including promising early results within the cardiac surgical community.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Sex: both; male and female
* Age (21-60) years old.
* American society of anesthesiology (ASA): II and III.
* Body mass index (BMI) >35 kg/m2
* Elective cardiac surgeries requiring median sternotomy.
* Accepted mental state of the patient.
* Non-smoker or ex-smoker for more than one month.
* Optimal preoperative glycemic control, defined by a hemoglobin A1c level less than 6.5%.

Exclusion Criteria:

* Patient refusal and lack of informed consent.
* Emergency or non-median sternotomy surgery.
* History of allergy to local anesthetics (lidocaine or bupivicaine).
* Coexisting hematologic disorders or malnourished patient.
* Pre-existing major organ dysfunction including hepatic or renal failure, and left ventricular ejection fraction <30%
* Peripheral neuropathy.
* Pregnancy.
* Patients with a diagnosis of cognitive impairment.
* Significant psychiatric illnesses including schizophrenia, bipolar disorder, uncontrolled anxiety, or depression.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
change in assessment of postoperative pain will be assessed by visual analogue scale (VAS) scale | at 1, 2, 3, 4, 8, 12, 16, 20 and 24 hours postoperatively
  scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.
The first requirement for analgesia: | within 24 hour postoperative
  The time from injection of LA to patient first request of analgesia

SECONDARY OUTCOMES:
Total amount of morphine consumed | within 24 hour postoperative
  Total amount of morphine given to each patient
Extubation time | within 24 hour postoperative
  Time from ICU admission to the time the endotracheal tube will be pulled out
ICU stay | within 24 hour postoperative
  Time from ICU admission to time of discharge to ward

CONTACTS AND LOCATIONS:
Overall Officials: Howaida A Kamal, MD, Study Director — faculty of medicine, Zagazig university, Egypt
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Fleming IO, Garratt C, Guha R, Desai J, Chaubey S, Wang Y, Leonard S, Kunst G. Aggregation of Marginal Gains in Cardiac Surgery: Feasibility of a Perioperative Care Bundle for Enhanced Recovery in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):665-70. doi: 10.1053/j.jvca.2016.01.017. Epub 2016 Jan 16. PMID 27321791
- [Background] Grant MC, Isada T, Ruzankin P, Whitman G, Lawton JS, Dodd-O J, Barodka V; Johns Hopkins Enhanced Recovery Program for the Cardiac Surgery Working Group. Results from an enhanced recovery program for cardiac surgery. J Thorac Cardiovasc Surg. 2020 Apr;159(4):1393-1402.e7. doi: 10.1016/j.jtcvs.2019.05.035. Epub 2019 Jun 7. PMID 31279510
- [Background] Li M, Zhang J, Gan TJ, Qin G, Wang L, Zhu M, Zhang Z, Pan Y, Ye Z, Zhang F, Chen X, Lin G, Huang L, Luo W, Guo Q, Wang E. Enhanced recovery after surgery pathway for patients undergoing cardiac surgery: a randomized clinical trial. Eur J Cardiothorac Surg. 2018 Sep 1;54(3):491-497. doi: 10.1093/ejcts/ezy100. PMID 29514224
- [Background] Ueshima H, Takeda Y, Ishikawa S, Otake H. RETRACTED: Ultrasound-guided transversus thoracic muscle plane block: a cadaveric study of the spread of injectate. J Clin Anesth. 2015 Dec;27(8):696. doi: 10.1016/j.jclinane.2015.05.013. Epub 2015 Jul 3. No abstract available. PMID 26144912 (Retraction: PMID 35396105 J Clin Anesth. 2022 Aug;79:110781)
- [Background] Barr AM, Tutungi E, Almeida AA. Parasternal intercostal block with ropivacaine for pain management after cardiac surgery: a double-blind, randomized, controlled trial. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):547-53. doi: 10.1053/j.jvca.2006.09.003. Epub 2006 Dec 22. PMID 17678782